CLINICAL TRIAL: NCT04620382
Title: Effect of Midodrine vs Abdominal Compression on Cardiovascular Risk Markers in Autonomic Failure Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Luis E Okamoto, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 201649; 1R01HL144568-01A1 (NIH)
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Neurogenic Orthostatic Hypotension; Autonomic Failure; Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease
Keywords: midodrine; abdominal binder; splanchnic circulation; arterial stiffness
MeSH Terms: conditions — Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease | interventions — Midodrine; Sugars

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, crossover
Who Masked: Participant
Masking Description: placebo pill and sham abdominal compression will be used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Midodrine (Active Comparator): Single oral dose of midodrine (5-10mg) combined with sham abdominal compression
  Interventions: Drug: Midodrine; Device: sham compression
- Abdominal Compression (Experimental): Abdominal compression (up to 40 mmHg) combined with a placebo pill
  Interventions: Drug: Placebo pill; Device: Abdominal compression

INTERVENTIONS:
Drug: Midodrine — Midodrine 5-10 mg, single oral dose
  Arms: Midodrine
Drug: Placebo pill — single oral dose
  Other Names: sugar pill
  Arms: Abdominal Compression
Device: Abdominal compression — abdominal compression up to 40 mmHg during head-up tilt
  Arms: Abdominal Compression
Device: sham compression — Sham abdominal compression during head-up tilt
  Arms: Midodrine

SUMMARY:
The purpose of this study is to learn more about the effects of abdominal compression and the medication midodrine, two interventions used for the treatment of orthostatic hypotension (low blood pressure on standing), on hemodynamic markers of cardiovascular risk. The study will be conducted at the Vanderbilt University Medical Center and consists of a screening and 2 testing days, one with abdominal compression and one with midodrine. The total length of the study will be about 5 days.

DETAILED DESCRIPTION:
The study includes up to 5 days spent in the Vanderbilt University Medical Center, at least one day of screening tests, followed by 2 study days.

Screening tests include a physical examination and history, routine safety laboratory assessments, and testing of the autonomic nervous system. Medications affecting blood pressure and the autonomic nervous system such as pressor medications will be withdrawn for at least 5 half-lives before studies, except for fludrocortisone. Other medications will be held constant throughout the study.

Eligible participants will then be studied on two separate days in random order: one day with midodrine combined with sham abdominal compression, and one day with abdominal compression combined with a placebo pill.

On each study day, participants will be instrumented to measure blood pressure, heart rate, hemodynamic parameters, segmental impedance, and markers of cardiovascular risk. A baseline tilt table test will be performed to obtain supine and upright baseline measurements, including the assessment of orthostatic symptoms. Participants will then receive a single oral dose of placebo or midodrine, and a deflated binder will be placed around the abdomen. Thirty to sixty minutes later, a second tilt table test will be done with sham or active abdominal compression. Outcome measurements will be repeated in the supine and upright positions. At the end of the second tilt table test, the investigators may also assess splanchnic venous capacitance.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years, with autonomic failure including pure autonomic failure, multiple system atrophy and Parkinson disease.
* Neurogenic orthostatic hypotension, defined as a ≥20-mmHg decrease in SBP within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes.
* Patients who are willing and able to provide informed consent

Exclusion Criteria:

* Pregnancy.
* Patients with any contraindication or intolerant to abdominal compression including history of aortic aneurysms, thoracic, abdominal or pelvic surgery within 6 months of study participation; symptomatic abdominal or inguinal hernias; severe gastrointestinal reflux; recent fractures or fissures of ribs, thoracic or lumbar spine; medical devices implanted on the abdominal wall or abdomen that would interfere with the abdominal compression.
* Pre-existing sustained supine hypertension ≥180/110mmHg
* Bedridden patients or those who are unable to stand due to motor impairment or severe OH.
* Patients who cannot tolerate the medication withdrawal, defined as those who are unable to stand for at least one minute after the medication withdrawal period or those with sustained supine hypertension ≥180/110mmHg.
* Clinically unstable coronary artery disease, or major cardiovascular or neurological event in the past 6 months.
* Clinically significant pulmonary, renal, hematopoietic, hepatic disease, or other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental, or laboratory testing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic markers of cardiovascular risk | 1 hour post-intervention tilt table test
  augmentation index, central blood pressure, pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Luis Okamoto, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04620382/ICF_000.pdf